CLINICAL TRIAL: NCT06006481
Title: Comparison of Physiotherapists Working in Different Fields in Terms of Occupational Satisfaction, Burnout, Musculoskeletal System Problems and the Strategies They Developed to Cope With it.
Brief Title: Musculoskeletal Problems and Strategies Developed by Physiotherapists to Cope With Them
Status: Completed | Type: Observational
Sponsor: Uskudar University (Other)
Responsible Party: Principal Investigator, Dr. Öğr. Üyesi Ömer Şevgin, Asst. Prof. Dr., Uskudar University
Other Study IDs: Uskudar57
Record Dates: First submitted 2023-08-17; First posted 2023-08-23 (Actual); Last update posted 2024-06-17 (Actual); Status verified 2024-06

CONDITIONS: Occupational Diseases; Muscle Pain
Keywords: physiotherapist; burnout; professional satisfaction
MeSH Terms: conditions — Occupational Diseases; Myalgia; Burnout, Psychological | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- 1.group: patient area in the children's area
  Interventions: Other: Survey
- 2.group: patient area in the field of orthopedics and athletes
  Interventions: Other: Survey
- 3.group: patient area in neurology and intensive care
  Interventions: Other: Survey
- 4.group: general group receiving patients in many fields
  Interventions: Other: Survey
- 5.group: physiotherapists working in public health
  Interventions: Other: Survey

INTERVENTIONS:
Other: Survey — Extended Nordic Musculoskeletal Questionnaire Pain Management Inventory Maslach Burnout Scale Vocational Satisfaction Scale

SUMMARY:
The aim of this study is to investigate whether there is a difference in areas such as occupational musculoskeletal injuries and strategies developed by physiotherapists working in different fields, burnout and occupational satisfaction.

DETAILED DESCRIPTION:
This study is a descriptive, cross-sectional online survey study. In this study, it is aimed to reach people who have graduated from the Physiotherapy and Rehabilitation Departments of the Faculties of Health Sciences or the Physical Therapy and Rehabilitation Schools of universities in Turkey, which provide education for 4 years and have the title of "physiotherapist". Physiotherapists will be divided into 5 groups according to the fields they work. Group 1 is only pediatric patients, Group 2 is orthopedics and sportsman, Group 3 is neurology and intensive care, Group 4 is general group that receives patients in many fields, and Group 5 is physiotherapists working in the field of public health. planned to occur. Before starting the study, the participants will be asked to fill in the Volunteer and Consent Form that they voluntarily participated in, and then they will be asked to fill out the Personal Information Form, the Extended Nordic Musculoskeletal System Questionnaire, the Pain Coping Inventory, the Maslach Burnout Scale, and the Vocational Satisfaction Scale prepared by us. According to the results obtained, 5 different groups will be compared among themselves by the determined parameters. The surveys to be used will be uploaded to the Google Forms database. Then, the participants will be asked to participate in the study by being reached via online media such as e-mail, mobile phone applications , social media.

ELIGIBILITY:
Inclusion Criteria:

* Volunteering to participate in the study
* Being a physiotherapist
* Having completed at least 1 year in the profession and continuing an active working life
* Being between the ages of 21 and 60

Exclusion Criteria:

* Not having completed 1 year in the profession
* Having any systemic disease

Ages: 21 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: physiotherapists who have been actively working for more than a year
Sampling Method: Non-Probability Sample
Enrollment: 255 (Actual)
Dates: Start 2023-09-01 (Actual); Primary Completion 2023-09-15 (Actual); Study Completion 2023-12-01 (Actual)

PRIMARY OUTCOMES:
Extended Nordic Musculoskeletal Questionnaire | 2 days
  It is a scale used to determine the extent of pain in the musculoskeletal system. The purpose of this questionnaire is to identify and compare pain and complaints in parts of the body. There is an image showing the 9 parts of the body included in the questionnaire. These body parts; neck, shoulders, back, elbows, hands, waist, hips, knees and feet. The respondents are asked whether they have experienced problems such as pain and discomfort in their body parts in the last 12 months, in the last 4 weeks, and on the day of the assessment, and they are asked to mark this as yes or no.
Maslach Burnout Scale | 2 days
  The scale consists of 22 questions in total. A 5-point Likert scale is used to answer the questions. There are options such as 0- Never, 1- Rarely, 2- Sometimes, 3- Often, 4- Always. Volunteers are asked to tick the appropriate option for each question. The scale has 3 sub-categories. There are 9 items for the emotional exhaustion section, 5 items for the depersonalization section, and 8 items for the personal achievement section. People with high burnout levels are expected to have high scores on the emotional exhaustion section and depersonalization section, and low personal achievement scores. The scores that can be obtained from the subscales range from 0-36 for emotional exhaustion, 0-20 for depersonalization, and 0-32 for personal achievement.
Vocational Satisfaction Scale | 2 days
  There are 20 questions in the scale. A five-point Likert-type rating scale was used for these questions. These ratings are 1. Always, 2. Often, 3. Sometimes, 4. Rarely, 5. Never. Items 1, 2, 3, 5, 6, 7, 8, 12, 13, 15, 16, 17, 18, 20 in the questions "5: Always, 4: Often, 3: Occasionally, 2: Rarely, 1: Never", while the items 4, 9, 10, 11, 14, 19, which make up the Negative items, are reversed; It should be scored as 1: Always, 2: Often, 3: Sometimes, 4: Rarely, 5: Never.
Pain Coping Inventory | 2 days
  It is a scale developed to determine the behavioral and cognitive strategies used by people with chronic pain to cope with this situation. In the original form of the scale, active as pain transformation, distancing and demand reduction; There are six passive sub-dimensions: withdrawal, worry, and rest. There are 22 questions in the scale and evaluation is made according to the 4-point Likert type. The lowest score is between 1 (almost never) and the highest score 4 (very often).

CONTACTS AND LOCATIONS:
Overall Officials: Elif SANDIKÇI, Study Chair — Bahçeşehir University
Locations (1):
- Turkey, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hou FI, Wu YL, Li MH, Huang WY. Physiotherapist' job performance, impression management and organizational citizenship behaviors: An analysis of hierarchical linear modeling. PLoS One. 2021 May 21;16(5):e0251843. doi: 10.1371/journal.pone.0251843. eCollection 2021. PMID 34019557
- [Background] Bridgeman PJ, Bridgeman MB, Barone J. Burnout syndrome among healthcare professionals. Am J Health Syst Pharm. 2018 Feb 1;75(3):147-152. doi: 10.2146/ajhp170460. Epub 2017 Nov 28. No abstract available. PMID 29183877
- [Background] Wasoski RL. Stress, professional burnout and dentistry. J Okla Dent Assoc. 1995 Fall;86(2):28-30. PMID 9526243
- [Background] Mroczek B, Lubkowska W, Jarno W, Jaraczewska E, Mierzecki A. Occurrence and impact of back pain on the quality of life of healthcare workers. Ann Agric Environ Med. 2020 Mar 17;27(1):36-42. doi: 10.26444/aaem/115180. Epub 2019 Dec 30. PMID 32208577
- [Background] Marik TL, Roll SC. Effectiveness of Occupational Therapy Interventions for Musculoskeletal Shoulder Conditions: A Systematic Review. Am J Occup Ther. 2017 Jan/Feb;71(1):7101180020p1-7101180020p11. doi: 10.5014/ajot.2017.023127. PMID 28027039